CLINICAL TRIAL: NCT06031662
Title: Image-guided, Accelerated, Theta-burst Stimulation for the Treatment of Post-concussion Syndrome
Brief Title: Accelerated, Theta-burst Stimulation for the Treatment of Post-concussion Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Sean Michael Nestor, clinician-investigator and interventional psychiatrist, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 5821
Record Dates: First submitted 2023-06-20; First posted 2023-09-11 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Post Concussion Syndrome
MeSH Terms: conditions — Post-Concussion Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental)
  Interventions: Device: Intermittent Theta-Burst Stimulation
- Sham (Sham Comparator)
  Interventions: Device: Sham Intermittent Theta-Burst Stimulation

INTERVENTIONS:
Device: Intermittent Theta-Burst Stimulation — Accelerated course of left dlPFC iTBS, consisting of 600 pulses/session, 50 minutes intersession interval, 8 session/day for 5 days) at 90% resting MT
  Arms: Treatment
Device: Sham Intermittent Theta-Burst Stimulation — Magventure Active/Placebo B70 coil specifically designed for randomized clinical trials with TMS. This system uses electrodes placed on the scalp to provide stimulation mimicking the active treatment condition
  Arms: Sham

SUMMARY:
TMS has been safely and reliably delivered at the Harquail Centre for over 5 years, with a primary focus on conventional rTMS protocols for treatment-resistant depression. Recently, the investgator team has gained the capability to deliver sham-controlled intermittent theta-burst stimulation (iTBS) rTMS. Unlike conventional high frequency rTMS, which was used in the previous sham-controlled rTMS PCS pilot study, iTBS is a patterned form of stimulation that recapitulates endogenous activity patterns of neural circuits pairing gamma frequency (50Hz) burst pulses coupled in a theta frequency rhythm (5Hz).12 iTBS delivers 600 pulses in just over 3 minutes with similar or greater effects on neural plasticity compared to conventional rTMS (taking over 30-45 minutes) and similar tolerability and efficacy in trials of depression. Furthermore, novel accelerated iTBS protocols stimulating the left dorsolateral prefrontal cortex (dlPFC) over 8-10 treatments, 50 minutes apart over a 5 day interval has recently demonstrated robust efficacy in depression and received recent FDA approval. Thus, accelerated iTBS can be delivered in a single week of treatment compared to 6 weeks with conventional rTMS methods. Finally, the investigators recently acquired the technology to integrate MRI neuroimage-guided stimulation, which would allow to target specific brain regions/networks implicated in PCS at high spatial resolution. No studies to date have investigated image-guided accelerated iTBS rTMS for the treatment of PCS.

ELIGIBILITY:
Inclusion Criteria:

* Documented evidence of head trauma sufficiently severe to result in loss of consciousness, post-traumatic amnesia and/or acute altered mental status.
* At least three symptoms including headache, dizziness, fatigue, irritability, insomnia, memory difficulties, concentration difficulties, mood dysregulation.
* Onset of symptoms within 4 weeks following the head trauma.
* Age 18-60, inclusive.
* Persistence of PCS symptoms for at least 3 months but less than 12 months
* Able to provide informed consent and comply with the study protocol
* Patients will not be excluded solely on the basis of communication (i.e., non-English speaking) unless they have exclusion criteria that is the cause of the communication difficulties.

Exclusion Criteria:

* Evidence of major structural neuroimaging abnormalities (e.g., intracranial hemorrhage, skull fracture or a large intracranial lesion)
* History of prior rTMS therapy,
* Contraindications to MRI (e.g., pacemaker, metallic implants etc.).
* Ferromagnetic, non-removable metallic implants from above the clavicle with the exception of dental work.
* Active personal injury litigation
* History of seizure disorder, not including febrile seizures in childhood
* Substance dependence within the last 6 months
* Pregnant
* Currently taking more than lorazepam 2 mg daily (or benzodiazepine equivalent) or any dose of an anticonvulsant (due to the potential to reduce rTMS efficacy)
* Currently taking an antiepileptic medication
* Mild and major comorbid medical conditions (as determined by investigators - e.g., neurological diseases, uncontrolled hypertension or diabetes, malignancy)
* A major comorbid psychiatric disorder (as determined by investigators - e.g., schizophrenia or bipolar disorder) and/or psychosis at the time of study enrollment

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2023-10-31 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Rivermead Post Concussion Symptoms Questionnaire | Baseline, change from baseline to immediately before the first iTBS treatment
  RPQ, a validated measure of subjective global PCS symptoms.
Rivermead Post Concussion Symptoms Questionnaire | 5 days
  RPQ, a validated measure of subjective global PCS symptoms.
Rivermead Post Concussion Symptoms Questionnaire | 1 month post-treatment
  RPQ, a validated measure of subjective global PCS symptoms.

SECONDARY OUTCOMES:
Montgomery-Åsberg Depression Rating Scale | Baseline, post treatment day 5, and post treatment 1 month
  Montgomery-Åsberg Depression Rating Scale is a widely used clinician-rated measure of depressive severity
Repeatable Battery for the Assessment of Neuropsychological Status | Baseline and post treatment 1 month
  RBANS is a brief, individually administered battery to measure cognitive decline or improvement
The Behavior Rating Inventory of Executive Function | Baseline, post treatment day 5, and post treatment 1 month
  BRIEF-A is a standardized measure that captures views of an adult's executive functions or self-regulation in his or her everyday environment.
Headache Impact Test | Baseline and post treatment 1 month
  HIT is a tool used to measure the impact headaches have on your ability to function on the job, at school, at home and in social situations.

CONTACTS AND LOCATIONS:
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No